CLINICAL TRIAL: NCT00172783
Title: PPD Size and Mycobacteria Tuberculosis ELISPOT in Children Who Have Received BCG in Neonate Period
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 940201
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-06

CONDITIONS: Tuberculosis
Keywords: TB; PPD; ELISPOT; BCG
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
To investigate the size of PPD and TB specific ELISPOT among children between 3m/o and 15 y/o . Calculate the normal range of age specific PPD size in children who recieved BCG at new-born period.

DETAILED DESCRIPTION:
Sampling

1. Age under 3 year-old: a targeted population contains 500 children will be used for sampling of this group. This cohort were firstly enrolled for a trial of oral Rota vaccine since 2004. They will be followed up in the cohort up to 2006. Sixty children will be enrolled in the group younger than 1 year-old (1-2, 2-3 year-old, 20 children will be enrolled in each age group).
2. Age of 3 to 5 year-old, cases will be enrolled from volunteered students from kindergarden (3-4, 4-5, 5-6 year-old, 20 children will be enrolled in each age group)
3. Age of 6 to 15 year-old, cases will be enrolled from volunteered students from elementary school and junior high school ( 30 children will be enrolled in each age group). A total of 300 children will be enrolled from children between 6 year-old and 15 year-old.

3. A total of 460 children between the age of 3 month and 15 y/o will be enrolled.

Procedure of PPD test Children who fit the criteria will be given 0.1 ml of PPD (PPD RT23, 2 units) intradermally, in accordance with the guidelines recommended by WHO (17). The tuberculin for the tests is obtained from Denmark and is used throughout the country. PPD indurations will be read 48 to 72 h after administration at 90 degrees from the longest axis of the arm and recorded to the nearest millimeter. Indurations <=5 mm in diameter are classified as negative, those >5 but <=10 mm as doubtful and those >10 mm as positive according to previous consensus (2). All size of indurations will be recorded for further analysis other than arbiturary classification.

Procedure of ELISPOT assay to detect T cells specific for M. tuberculosis antigens 4 ml whole blood is collected in a heparinized tube first and are processed and scored by two scientists who had no access to personal identifiers or TST results within four hours after collection. We amplified the esat-6 gene from genomic DNA isolated from M bovis strain AN5 by PCR, and cloned it into plasmid vector pET21d (Novagen, Madison, WI, USA). Escherichia coli was transformed with this vector. Recombinant ESAT-6 was recovered from transformed E coli and purified by nickel-affinity chromatography. We did ex-vivo interferon-gamma ELISPOT assays, with 300 000 peripheral blood mononuclear cells per well (14,18). We used purified recombinant ESAT-6 and PPD, in addition to negative controls (no added antigen) and positive controls (phytohaemagglutinin). Positive ESAT-6 test wells were defined as containing at least ten spot-forming cells more than, and at least twice as many as, negative control wells-a detection threshold of one per 30 000 peripheral blood mononuclear cells. Assays were done and independently scored by two scientists who were unaware of exposure category and TST results of contacts. ELISPOT assay wells containing more than 300 spot-forming cells cannot be counted accurately because the spots coalesce. 300 cells per well (equivalent to 1000 cells per million peripheral blood mononuclear cells) was therefore taken as the upper limit for accuracy (15).

Exclusion and Follow-up steps Children who are found to have positive PPD test (>10 mm), have a PPD size in the range of 1st 2.5 percentile or having a positive ELISPOT result at the time of enrollment, will be closely followed up for clinical symptoms and signs of TB and necessary diagnostic workup will be done. If LTBI is highly suspected, prophylaxis will be initiated. Closed contact families and care-givers will be asked to take CXR for excluding active pulmonary TB.

Information collection at the enrollment Cross-sectional study of 160 children will be conducted. Children were examined and assessed for general health condition, BCG vaccination record, and BCG scar over L't arm (19). Possible TB exposure including elderly with chronic cough or unexplained prolonged febrile illness in house-hold contact, any contact history with documented open TB will be thoroughly evaluated. Children with suspicious immuno-compromised status, active lung disease or exposure history of TB will be excluded and follow-up will be done.

Biostatistic method Descriptive analysis will be used for size of PPD and result of ELISPOT. P value is calculated with student t test or Chi-square or Fisher exact test for statistic significance (Version 10.0, SPSS, SPSS Inc. Illinois) between different age group. 95%CI will be calculated for the purpose of cut off value of PPD size (except those with unexpected-found TB disease).

ELIGIBILITY:
Inclusion Criteria: A healthy child with the age between 3 month to 15 year, who has received BCG in the first month of life as schedule, without history of exposure of tuberculosis. -

Exclusion Criteria: Children not received his BCG within one month after birth, immunodeficiency, received steroid or immunosuppresant within 6 weeks, severe infection within 6 weeks, received life vaccine within 6 weeks

-

Ages: 3 Months to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 460
Dates: Start 2005-06; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Li-Ming Huang, MD, PHD, Study Chair — National Taiwan University Hospital, Pediatrics
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan